CLINICAL TRIAL: NCT05602220
Title: Heart Rate and Breathing Effects on Attention and Memory
Acronym: HeartBEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mara Mather, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UP-21-00357
Record Dates: First submitted 2022-09-06; First posted 2022-11-02 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Aging; Alzheimer Disease; Age-related Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain training and paced breathing to stimulate alertness (Experimental)
  Interventions: Behavioral: Brain training; Behavioral: Paced breathing
- Brain training and paced breathing to relax (Experimental)
  Interventions: Behavioral: Brain training; Behavioral: Paced breathing

INTERVENTIONS:
Behavioral: Brain training — Participants will play a few brain training games using an online interface each day. These games train attention, memory and other cognitive functions.
Behavioral: Paced breathing — After completing brain training, they will then immediately do one 15-minute session of paced breathing, followed by a second 15-min session of paced breathing later in the day. During the paced breathing sessions, participants will clip a pulse monitor to their ear lobe and try to inhale and exhale in synchrony with a ball that moves up and down on the screen. They will receive heart rate biofeedback regarding whether they are achieving their relaxation/alertness goal.

SUMMARY:
In the current study, we will examine how daily paced breathing affects plasma amyloid beta levels and the rate of learning in older adults. Healthy adults aged 50-70 who meet all eligibility criteria will be invited to this study. Participants will be randomly assigned to one of the two conditions: 1) Daily memory and attention training followed by a paced breathing protocol designed to increase relaxation or 2) Daily memory and attention training followed by a paced breathing protocol to increase alertness. Participants will be asked to complete pre and post intervention cognitive testing online, engage in 10 weeks of daily brain training (starting Week 2) and 9 weeks of paced breathing (starting Week 3) at home. They will also be asked to come in for lab visits on Weeks 2, 7 and 12 to provide blood and urine samples to assess amyloid beta levels and to complete magnetic resonance imaging scans to assess perivascular space volume.

ELIGIBILITY:
Inclusion Criteria:

* speak English fluently
* between the age of 50-70
* healthy adult who weighs at least 110 pounds
* non-pregnant and non-menstruating (for at least the past year)
* normal or corrected-to-normal vision and hearing
* have a home computer with a physical keyboard and have access to reliable internet
* have an email account that you check regularly
* have a phone that receives text messages
* willing to provide a blood sample and a urine sample at three lab visits
* willing to devote up to 60 minutes daily to the study for 12 weeks (in addition to lab visits)

Exclusion Criteria:

* have a disorder that would impede performing the breathing intervention (e.g., abnormal cardiac rhythm, heart disease including coronary artery disease, angina, and arrhythmia, cognitive impairment, dyspnea)
* regularly practicing any relaxation, biofeedback, or breathing technique (e.g., meditation) for more than an hour a week
* regularly played Lumosity games in the past 6 months
* participated in heart rate biofeedback studies in the USC Emotion & Cognition Lab
* have any conditions listed below that are not safe for MRI

  * Claustrophobia
  * Have worked as a machinist, metal worker, or in any profession or hobby grinding metal?
  * Have had an injury to the eye involving a metallic object (e.g., metallic slivers, shavings, or foreign body)
  * Cardiac pacemaker
  * Implanted cardiac defibrillator
  * Aneurysm clip or brain clip
  * Carotid artery vascular clamp
  * Neurostimulator
  * Insulin or infusion pump
  * Spinal fusion stimulator
  * Cochlear, otologic, ear tubes or ear implant
  * Prosthesis (eye/orbital, penile, etc.)
  * Implant held in place by a magnet
  * Heart valve prosthesis
  * Artificial limb or joint
  * Other implants in body or head
  * Electrodes (on body, head or brain)
  * Intravascular stents, filters
  * Shunt (spinal or intraventricular)
  * Vascular access port or catheters
  * IUD
  * Transdermal delivery system or other types of foil patches (e.g., Nitro, Nicotine, Birth control, etc.) that cannot be removed for MRI
  * Shrapnel, buckshot, or bullets
  * Tattooed eyeliner or eyebrows
  * Body piercing(s) that cannot be removed for MRI
  * Metal fragments (eye, head, ear, skin)
  * Internal pacing wires
  * Aortic clips
  * Metal or wire mesh implants
  * Wire sutures or surgical staples
  * Harrington rods (spine)
  * Bone/joint pin, screw, nail, wire, plate
  * Wig or toupee that cannot be removed for MRI
  * Hair implants that involve staples or metal
  * Hearing aid(s) that cannot be removed for MRI
  * Dentures or retainers that cannot be removed for MRI

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Nashiro K, Yoo HJ, Cho C, Kim AJ, Nasseri P, Min J, Dahl MJ, Mercer N, Choupan J, Choi P, Lee HRJ, Choi D, Alemu K, Herrera AY, Ng NF, Thayer JF, Mather M. Heart rate and breathing effects on attention and memory (HeartBEAM): study protocol for a randomized controlled trial in older adults. Trials. 2024 Mar 15;25(1):190. doi: 10.1186/s13063-024-07943-y. PMID 38491546

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 91 participants enrolled, 10 dropped after enrolling but before Week 1 home assessments, and an additional 19 dropped before condition assignment.
Period: Overall Study
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Started | 31 | 31
Completed | 29 | 31
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.77 (6.17) | 60.52 (5.42) | 60.15 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 16 | 18 | 34
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Amyloid Beta (Aβ) Levels
Description: We computed an aggregate Z-score based on plasma Aβ40 and Aβ42 levels (pg/mL). A Z-score of 0 represents the sample mean. Higher values indicate a greater level of plasma Aβ, which in cognitively normal individuals has been found to be associated with a higher risk of converting to Alzheimer's disease (Song et al., 2011). This score was compared across three time points: Week 2 (pre-intervention), Week 7 (mid-intervention), and Week 12 (post-intervention). We conducted a time (Week 2, 7, 12) × condition ANOVA to test for a time × condition interaction in plasma Aβ levels, assessing group differences in change over time.
Time Frame: Measured from blood draws at lab visits on Weeks 2, 7, and 12
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Number analyzed (Participants) | 27 | 31
Z-score
  Week 2 | 0.343 (0.161) | -0.371 (0.150)
  Week 7 | 0.381 (0.161) | -0.332 (0.151)
  Week 12 | 0.410 (0.161) | -0.387 (0.150)
Statistical Analysis 1: Comparison: Brain Training and Paced Breathing to Stimulate Alertness vs Brain Training and Paced Breathing to Relax; Test type: Superiority; p = 0.817, ANOVA; F test = 0.054

2. Primary Outcome: Change in Plasma Ab42/40 Ratio
Description: The plasma Aβ42/40 ratio was calculated by dividing the plasma Aβ42 concentration (pg/mL) by the plasma Aβ40 concentration (pg/mL) at each time point. We conducted a time (Week 2, 7, 12) × condition ANOVA to test for an interaction effect, using plasma Aβ42/40 ratio scores as the dependent variable to assess group differences over time. A higher Aβ42/40 ratio indicates a better outcome, reflecting greater brain clearance of Aβ.
Time Frame: Measured from blood draws at lab visits on Weeks 2, 7, and 12
Measure: Mean (Standard Error); unit: ratio of Aβ42 to Aβ40
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Number analyzed (Participants) | 27 | 31
ratio of Aβ42 to Aβ40
  Week 2 | .040 (.001) | .038 (.001)
  Week 7 | .041 (.001) | .039 (.001)
  Week 12 | .040 (.001) | .037 (.001)
Statistical Analysis 1: Comparison: Brain Training and Paced Breathing to Stimulate Alertness vs Brain Training and Paced Breathing to Relax; Test type: Superiority; p = 0.147, ANOVA; F test = 2.162

3. Secondary Outcome: Change in Brain Perivascular Space Volume
Description: We tested whether there were group differences in changes in perivascular space (PVS) volume. PVS volume was defined as the percentage of PVS volume relative to white matter volume in the centrum semiovale, our main region of interest.
Time Frame: Measured from magnetic resonance imaging completed at lab visits on Weeks 2, 7, and 12
Measure: Mean (Standard Deviation); unit: percentage of PVS volume
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Number analyzed (Participants) | 25 | 29
percentage of PVS volume
  Week 2 | 0.0077 (0.0034) | 0.0079 (0.0043)
  Week 7 | 0.0083 (0.0042) | 0.0088 (0.0052)
  Week 12 | 0.0092 (0.0054) | 0.0080 (0.0039)
Statistical Analysis 1: Comparison: Brain Training and Paced Breathing to Stimulate Alertness vs Brain Training and Paced Breathing to Relax; Test type: Superiority; p = 0.096, ANOVA; F test = 2.88

4. Secondary Outcome: Change in Hippocampal Volume
Description: We tested whether there were group differences in changes in hippocampal volume. We performed a two-way mixed ANCOVA on hippocampal volume, with condition as the between-subjects factor and time point (Week 2, 7, 12) as the within-subjects factor, controlling for intracranial volume as a covariate.
Time Frame: Measured from magnetic resonance imaging completed at lab visits on Weeks 2, 7, and 12
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Number analyzed (Participants) | 26 | 29
mm^2
  Week 2 | 7036 (105.0) | 7143 (99.2)
  Week 7 | 7038 (105.6) | 7124 (99.8)
  Week 12 | 7018 (103.1) | 7102 (97.4)
Statistical Analysis 1: Comparison: Brain Training and Paced Breathing to Stimulate Alertness vs Brain Training and Paced Breathing to Relax; Test type: Superiority; p = 0.640, ANCOVA; F test = 0.449

5. Secondary Outcome: Brain Training Performance on 12 Lumosity Games
Description: Participants completed 12 brain-training games on the Lumosity platform (https://www.lumosity.com/) targeting six cognitive domains: Attention, Flexibility, Language, Math, Memory, and Reasoning. Performance scores were expressed in arbitrary units, with minimum scores generally in the hundreds. The exact lower limits vary across games, and the upper limits differ substantially between games. Across all games, higher scores indicate better cognitive performance.
  For analyses, standardized performance scores (z-scores) were derived from the raw Lumosity game scores. Scores were standardized within each game across all participants; therefore, some values may appear negative, reflecting scores below the sample mean. A z-score of 0 represents the sample mean, with higher z-scores indicating better cognitive function. Standardized scores across games were combined using Partial Least Squares Correlation (PLSC) analyses.
Time Frame: Measured at pre-intervention during week 2 and at the end of the intervention during week 12
Measure: Mean (Standard Deviation); unit: Z-scores
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
Number analyzed (Participants) | 29 | 31
Z-scores
  baseline performance (bin1) | -2.9144 (1.3024) | -2.9242 (1.1478)
  final performance (bin 10) | 1.5021 (2.2580) | 1.4551 (1.9558)
Statistical Analysis 1: Comparison: Brain Training and Paced Breathing to Stimulate Alertness vs Brain Training and Paced Breathing to Relax; Test type: Superiority — Linear mixed-effects model fit to participants' latent performance scores across 10 time bins. Comparison of performance changes over time between groups; p = 0.997, Mixed Models Analysis; beta parameter = 0.0001419, 95% CI 2-sided [-0.072164 to 0.072448], Standard Error of Mean 0.036816

6. Other Pre Specified Outcome: Change in Plasma pTau-181/Tau Ratio
Description: We will conduct a time (Week 2, 7, 12) X condition ANOVA to test for a time X condition interaction with plasma pTau-181/tau ratio as the dependent variable (to assess group differences in change).
Time Frame: Measured from blood draws at lab visits on Weeks 2, 7, and 12
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Urine Ab42
Description: We will conduct a time (Week 2, 7, 12) X condition ANOVA to test for a time X condition interaction with urine Ab42 as the dependent variable (to assess group differences in change).
Time Frame: Measured from urine samples at lab visits on Weeks 2, 7, and 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Brain Training and Paced Breathing to Stimulate Alertness | Brain Training and Paced Breathing to Relax
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 3/31 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brain Training and Paced Breathing to Stimulate Alertness (N=31) | Brain Training and Paced Breathing to Relax (N=31)
bruising following a blood draw (Blood and lymphatic system disorders) | 2 | 2 — Four participants reported experiencing more bruising than usual following their blood draw. However, during follow-up, all participants indicated they were feeling fine and that the bruising was resolving.
light-headedness during home practice (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — One participant reported experiencing nausea and light-headedness during their daily breathing practices. A researcher advised them to take soft shallow breaths instead of deep breathing, which alleviated the symptoms.
Discomfort during MRI due to body size (General disorders) | 1 | 0 — Participant experienced discomfort due to body size in MRI scanner. The bed got stuck, causing a brief delay. Staff provided support, and the participant was safely removed. Follow-up confirmed no lasting symptoms or injuries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05602220/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05602220/SAP_001.pdf